CLINICAL TRIAL: NCT03574727
Title: The Management of Abdominal Cutaneous Nerve Entrapment Syndrome
Brief Title: Abdominal Cutaneous Nerve Entrapment Syndrome
Acronym: ACNES
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017AN003
Record Dates: First submitted 2018-06-20; First posted 2018-07-02 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Abdominal Pain; Abdominal Cutaneous Nerve Entrapment Syndrome
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Injection to or release of anterior cutaneous nerves — Patients who have undergone at least one injection to the nerves

SUMMARY:
Nerve entrapment as a cause of chronic abdominal pain is frequently overlooked. A series of nerves pass through the muscles of the abdomen before reaching the skin to carry sensations. They can get trapped within the muscles leading to severe pain resulting in a condition known as Abdominal Cutaneous Nerve Entrapment Syndrome (ACNES). ACNES affects between 10-30% of patients with chronic abdominal wall pain. A definitive diagnosis of ACNES is obtained by anaesthetising these nerves. Initial management includes education and avoidance of known triggers. It is common practice to inject steroid with local anaesthetic during the diagnostic injections itself to prolong pain relief. Like other nerve entrapment conditions, this is also refractory to medical treatment. Hence repeated injections and nerve entrapment release surgery are commonly carried out.

In Aberdeen, a number of patients have been treated for this condition. A cohort of patients have benefitted with injection alone while recurrence has been noted in patients who have undergone surgery. This project aims to gain more understanding about the clinical course of patients with suspected ACNES by evaluation of the clinic progress.

DETAILED DESCRIPTION:
This is a cross-sectional survey, best suited to evaluate the effect of treatments. Potential participants will be identified from a list of patients who have attended the pain clinic at Aberdeen Royal Infirmary for chronic abdominal wall pain.

These patients will be invited to participate in the study via posted letter. The letter will include a participant information sheet detailing who is running the study, what the purpose of the study is, what participating in the study requires of a patient and how their information will be used.

Patients who wish to participate will return a note of interest, included within the participant information pack, and will then be invited to attend an outpatient clinic in the Aberdeen Health Care and Community Village. Informed consent will be obtained. The questionnaire will be distributed. It is estimated that the questionnaire will take approximately 15 minutes to complete. Each completed questionnaire will be reviewed immediately by a member of the research team to ensure all relevant sections have been completed. Following completion of the questionnaire, patients will be allowed to leave. It is not anticipated that participants will need to be contacted after submitting their completed questionnaire. Participants who explicit express the need for further pain management will be referred to NHS Grampian pain clinic.

A response from potential participants will be awaited for 4 weeks. In the event of no response, a maximum of 2 written reminders 4 weeks apart will be sent along with participant information pack.

The questionnaires have previously been validated for use in neuropathic pain, and the outcomes of the questionnaire are consistent with those recommended by the 2008 Initiative on Methods, Measurement and Pain Assessment in Clinical Trials (IMMPACT) publication. 17

The questionnaire will consist of four main sections: baseline demographic details, a detailed pain history prior to surgery, including questions from the Brief Pain Inventory, 18 open-ended questions to explore the patient's opinions of both the operation and their health status since and, finally, an overall picture of health using the European Quality of Life-5 Dimensions (EQ-5D) Score 19 and patient global impression of change scale. 20

In order to compare pain both before and after surgery, participants will be asked to complete these sections twice, focusing on their previous health state and their current health.

Since pain scores are not routinely collected and all patients will be seen after surgery, pre-operative pain scores will be retrospective.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for inclusion, all patients must:

* Be aged 16 or over
* Be able to understand English
* Be able to give informed consent
* Be able to report on their health and pain status (neurologically stable)
* Should have undergone either injection or surgery for suspected ACNES

Exclusion Criteria:

Patients will be excluded if they:

* Are not able to understand what is required of them
* Are not able to give informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Potential participants will be identified from the hospital electronic booking system.
  A list of patients between January 2010 and December 2015 and had injection for chronic abdominal wall pain will be invited for the study.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-09-19 (Actual)

PRIMARY OUTCOMES:
Success rate of intervention | 3 months
  An intervention either injection or surgery is classed as success when there is either a 2 point difference in the average pain scores pre and post intervention or more than 30% improvement as rated by the participant in the Brief Pain Inventory used for evaluating the pain baseline and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Saravanakumar Kanakarajan, MD, Principal Investigator — NHS Grampian
Locations (1):
- Aberdeen Royal Infirmary, Aberdeen, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kanakarajan S, Dharmavaram S, Tadros A, Pushparaj H, Rose A. Abdominal cutaneous nerve entrapment syndrome: A cross sectional survey of treatment outcomes. Br J Pain. 2022 Oct;16(5):538-545. doi: 10.1177/20494637221101719. Epub 2022 May 20. PMID 36389004
- See also: National Library of Medicine — https://pubmed.ncbi.nlm.nih.gov/36389004/